CLINICAL TRIAL: NCT05863975
Title: Therapeutic Effect of Topical Estrogen and Human Interferon Alpha 2b Vaginal Effervescent Capsules in Perimenopausal and Postmenopausal Women With High-risk HPV Infection
Brief Title: Treatment of HPV Infection in Perimenopausal and Postmenopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 49557358-X
Record Dates: First submitted 2023-03-26; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: HPV Infection
Keywords: Perimenopause; postmenopausal; HPV infection; treatment
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interferon group (Experimental): Vaginal placement of human interferon alpha 2b vaginal effervescent capsules, one pill a day daily, 10 days, for a course of treatment, a total of 3 courses
  Interventions: Drug: Human interferon alpha 2b vaginal Effervescent capsules
- Promestriene group (Experimental): promestriene cream vaginal medication, once a day, 1g each time, 10 days, for a course of treatment, a total of 3 courses of treatment
  Interventions: Drug: Human interferon alpha 2b vaginal Effervescent capsules
- Interferon + promestriene combination group (Experimental): given one human interferon alpha 2b vaginal effervescent capsule vaginal placement + promestriene cream 1g vaginal medication, once a day, for 10 days, for a course of 1, 3 courses of continuous use.
  Interventions: Drug: Human interferon alpha 2b vaginal Effervescent capsules

INTERVENTIONS:
Drug: Human interferon alpha 2b vaginal Effervescent capsules — ①Interferon group: human interferon alpha 2b vaginal effervescent capsule vaginal medication. ② Promestriene group: promestriene cream vaginal medication. ③Interferon + promestriene combination group: two drugs were given in combination.
  Other Names: Promestriene cream; Human interferon alpha 2b vaginal Effervescent capsules+Proestradiene cream

SUMMARY:
A randomized controlled study was conducted to determine the effects of vaginal estrogen and human interferon alpha 2b vaginal effervescent capsules on vaginal microecology in perimenopausal and postmenopausal women. To determine whether there is a synergistic effect between the two in the treatment of HPV infection in perimenopausal and postmenopausal women. To observe the effects of two drugs alone and combined on the vaginal immune environment of patients.

DETAILED DESCRIPTION:
After pre-enrollment screening, patients who met the inclusion criteria signed informed consent and were divided into interferon group, promestriene group and interferon + promestriene combination group according to the randomized controlled number table.

① Interferon group: human interferon alpha 2b vaginal effervescent capsules were given vaginal medication, one capsule a day for 10 days, for a course of treatment, a total of 3 courses of treatment. ② Promestriene group: Promestriene cream vaginal medication, once a day, 0.1g each time, 10 days, for a course of treatment, a total of 3 courses of treatment. ③Interferon + promestriene combination group: interferon 1 grain + promestriene cream 0.1g, vaginal medication, once a day, continuous use for 10 days, for a course of treatment, continuous use of 3 courses of treatment. Vaginal secretions were collected before treatment and one week after treatment to detect vaginal microecology. Flow cytometry was used to detect the proportion of immune cells in vaginal secretion. ELISA was used to detect immune-related cytokines (IFN-γ, TNF-α, IL-2, IL-4, IL-6, IL-10) in vaginal secretions.

HPV was reviewed at 1 month and 1 year after drug cessation.

ELIGIBILITY:
Inclusion Criteria:

* The age of 45-65 years (inclusive);

  * HPV test indicates positive cervical and vaginal high-risk HPV;

    * Cervical HSIL was excluded according to the 2015 US Transitional Clinical Guidelines for Cervical Cancer Screening.

      * Patients with high-grade cervical intraepithelial lesions, who have undergone cervical conotomy or have undergone total or subtotal hysterectomy in the past, and HPV tests indicate high-risk cervical and vaginal HPV infection;

        * If the combination of clear vaginal inflammation, symptomatic treatment is needed, then the group test;

          * If the patients were complicated with abnormal uterine bleeding or postmenstrual bleeding, the reproductive system tumor should be excluded and cured, and then the patients were re-enrolled.

            ⑦ Volunteer to participate in clinical studies and sign informed consent.

Exclusion Criteria:

* Allergic to human interferon alpha 2b vaginal effervescent capsules or prolestrene cream;

  * Pregnant or lactating patients;

    * Patients with abnormal vaginal bleeding without clear cause;

      ④Patients with cervical high-grade intraepithelial lesions, gynecological malignancies, serious heart, brain, kidney, immune, blood and other systems and psychiatric neuropsychological diseases;

      ⑤Patients with consciousness disorder and communication disorder can not cooperate with the experiment;

      ⑥ Patients considered unsuitable or refused to participate in this clinical trial.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV negative conversion rate | 1 month and 1 year after drug discontinuation
  Number of cases of HPV negative conversion after medication/total cases ×100%

SECONDARY OUTCOMES:
Vaginal microecological improvement | 1 week after drug discontinuation
  Concentration and diversity of vaginal microflora after drug treatment